CLINICAL TRIAL: NCT02619344
Title: Endothelial Dysfunction and Selenium Status in Children With Acute Systemic Inflammatory
Brief Title: Endothelial Dysfunction and Selenium Status in Children With Acute Systemic Inflammatory Response
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Emilio Lopes Junior, post graduate, Federal University of São Paulo
Other Study IDs: Endothelium
Record Dates: First submitted 2015-08-03; First posted 2015-12-02 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Endothelial Dysfunction; Regulation of Acute Inflammatory Response; Selenium Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall hypotheses of this project is that severe sepsis is associated with endothelial dysfunction in pediatric patients and that selenium deficiency is associated with changes in biological markers of endothelial dysfunction and that these changes, in turn, are associated with worse clinical prognosis.

DETAILED DESCRIPTION:
Background: Oxidative stress occurs during shock as a result of granulocytes and endothelial cell activation. Higher intensity of endothelial activation is associated with unfavorable outcomes. Selenium is an essential trace element that plays a key role in the antioxidant defenses and whose plasma concentrations have been low in critically ill patients. There are no clinical studies, especially in pediatric patients that consider the roles of selenium and nutritional status in the modulation of endothelial adaptive response during the inflammatory response secondary to shock. The investigators hypothesize that selenium deficiency is associated with changes in biological markers of endothelial dysfunction and that these changes, in turn, are associated with worse clinical prognosis. Objectives: 1) to investigate the association between selenium (Se) status and the endothelial activation in children during acute systemic inflammatory response and 2) to investigate whether the intensity of endothelial activation can predict the clinical outcome in children with systemic inflammatory response.

Methodology: prospective, observational study in children admitted to an intensive care unit (ICU) with systemic inflammatory response. The primary outcome will be 'intensity endothelial activation' which will be defined based on biological markers (SE-selectin, soluble intercellular molecule 1 of Vascular Cell adhesion Molecule and soluble adhesion-1). The association between the state of Se (anthropometric measurements, blood levels of selenium and erythrocyte glutathione peroxidase, selenoprotein P activity) and this outcome will be investigated in a multiple logistic model considering age, gender, primary diagnosis, prognostic scores and clinical characteristics. The secondary outcome will be 'clinical prognosis' which will be defined based on 'organ dysfunction' (creatinine level, platelets level and arterial hypotension), infectious complications during the staying in ICU and death up to 28 days. In this step the explanatory variables will be the same used in the first analyse plus to 'intensity of endothelial activation'. Participants will be followed for the duration of ICU/Hospital stay, an expected average of 28 days. Particularly, biological markers of endothelial activation will be evaluated in three different times: at baseline and on days 3 and 5 ICU. Expected results: if the study hypotheses are correct, they may justify the analysis of biomarkers of endothelial activation in medical practice and in future studies assessing the benefits of selenium supplementation in critical illness.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to an intensive care unit with systemic inflammatory response

Exclusion Criteria:

* Blood transfusion
* Chronic disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children admitted to an intensive care unit (ICU) with systemic inflammatory response.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
association between selenium status and the endothelial activation | 30/06/2016 (up to 2 years)
  To investigate the association between selenium status and the endothelial activation in children during acute systemic inflammatory response.

SECONDARY OUTCOMES:
Endothelial activation and clinical outcome in children with SIRS | 30/06/2016 (up to 2 years)
  To investigate whether the intensity of endothelial activation can predict the clinical outcome in children with systemic inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Heitor Pons Leite, professor, Study Director — Federal University of São Paulo
Locations (1):
- Emílio Lopes Junior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651